CLINICAL TRIAL: NCT02500381
Title: A Double-Blind, Placebo-Controlled, Multi-Center Study With an Open-Label Extension to Evaluate the Efficacy and Safety of SRP-4045 and SRP-4053 in Patients With Duchenne Muscular Dystrophy
Brief Title: Study of SRP-4045 (Casimersen) and SRP-4053 (Golodirsen) in Participants With Duchenne Muscular Dystrophy (DMD)
Acronym: ESSENCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4045-301; 2015-002069-52 (EudraCT Number); 2024-514698-23-00 (Other: CTIS Number)
Record Dates: First submitted 2015-07-14; First posted 2015-07-16 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; Exon Skipping; DMD; Exon 53; Exon 45; Ambulatory; Pediatric; Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — casimersen; golodirsen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 is double-blind and randomized; Part 2 is open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SRP-4045 (Experimental): Participants amenable to exon 45 skipping will receive SRP-4045 IV infusions, weekly, at 30 mg/kg for up to 96 weeks in the double-blinded period. This will be followed by an open-label extension period in which all participants will receive open-label active treatment of SRP-4045 at 30 mg/kg/week IV infusions for 48 weeks (up to Week 144 in the study).
  Interventions: Drug: SRP-4045
- SRP-4053 (Experimental): Participants amenable to exon 53 skipping will receive SRP-4053 IV infusions, weekly, at 30 mg/kg for up to 96 weeks in the double-blinded period. This will be followed by an open-label extension period in which all participants will receive open-label active treatment of SRP-4053 at 30 mg/kg/week IV infusions for 48 weeks (up to Week 144 in the study).
  Interventions: Drug: SRP-4053
- Placebo followed by SRP-4045 or SRP-4053 (Placebo Comparator): Participants amenable to exon 45 or 53 skipping will receive SRP-4045 or SRP-4053 placebo-matching IV infusions, weekly, at 30 mg/kg for up to 96 weeks in the double-blinded period. This will be followed by an open-label extension period in which all participants will receive open-label active treatment of SRP-4045 or SRP-4053 at 30 mg/kg/week IV infusions for 48 weeks (up to Week 144 in the study).
  Interventions: Drug: SRP-4045; Drug: SRP-4053; Drug: Placebo

INTERVENTIONS:
Drug: SRP-4045 — SRP-4045 solution for IV infusion
  Other Names: Casimersen; AMONDYS 45
  Arms: Placebo followed by SRP-4045 or SRP-4053; SRP-4045
Drug: SRP-4053 — SRP-4053 solution for IV infusion
  Other Names: Golodirsen; VYONDYS 53
  Arms: Placebo followed by SRP-4045 or SRP-4053; SRP-4053
Drug: Placebo — SRP-4045 or SRP-4053 placebo-matching solution for IV infusion
  Arms: Placebo followed by SRP-4045 or SRP-4053

SUMMARY:
The main objective of this study is to evaluate the efficacy of SRP-4045 (casimersen) and SRP-4053 (golodirsen) compared to placebo in participants with DMD with out-of-frame deletion mutations amenable to skipping exon 45 and exon 53, respectively.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, multi-center study to evaluate the efficacy and safety of SRP-4045 and SRP-4053. Eligible participants with out-of-frame deletion mutations amenable to exon 45 or 53 skipping will be randomized to receive once weekly intravenous (IV) infusions of 30 milligrams/kilograms (mg/kg) SRP-4045 or 30 mg/kg SRP-4053 respectively (combined-active group) or placebo for up to 96 weeks (the placebo-controlled period of the trial). This will be followed by an open-label extension period in which all participants will receive open-label active treatment for 48 weeks (up to Week 144 of study).

The study will enroll approximately 222 participants. Twice as many participants will be randomized to receive active treatment as will receive placebo (2:1 randomization).

Clinical efficacy will be assessed at regularly scheduled study visits, including functional tests, such as the 6-minute walk test (6MWT). All participants will undergo a muscle biopsy at baseline and a second muscle biopsy either at Week 48 or Week 96.

Safety will be assessed through the collection of adverse events (AEs), laboratory tests, electrocardiograms (ECGs), echocardiograms (ECHOs), vital signs, and physical examinations throughout the study.

Blood samples will be taken periodically throughout the study to assess the pharmacokinetics of both drugs.

ELIGIBILITY:
Inclusion Criteria:

* Genotypically confirmed DMD, with genetic deletion amenable to exon 45 or exon 53 skipping
* Stable dose of oral corticosteroids for at least 24 weeks prior to Week 1, and the dose is expected to remain constant throughout the study (except for modifications to accommodate changes in weight).
* Intact right and left biceps brachii muscles or 2 alternative upper arm muscle groups
* Mean 6MWT ≥300 meters and ≤450 meters
* Stable pulmonary function: forced vital capacity (FVC) ≥50% predicted

Exclusion Criteria:

* Treatment with gene therapy at any time
* Previous treatment with SMT C1100 within 1 week prior to Week 1 and previous treatment with PRO045 (BMN 045), PRO053 (BMN 053), or PRO051 (BMN 051) within 24 weeks prior to Week 1
* Current or previous treatment with any other experimental treatment within 12 weeks prior to Week 1
* Major surgery within 3 months prior to Week 1
* Presence of other clinically significant illness
* Other inclusion/exclusion criteria may apply.

Ages: 6 Years to 13 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 228 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2025-10-16 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in the 4-Step Ascend Velocity at Week 96 | Baseline, Week 96

SECONDARY OUTCOMES:
Change from Baseline in the Total Distance Walked During 6MWT at Week 96 | Baseline, Week 96
Change from Baseline in Rise from Floor Velocity at Week 96 | Baseline, Week 96
Change From Baseline in the 4-Step Ascend Velocity at Week 144 | Baseline, Week 144
Change From Baseline in Total Distance Walked During the 10-meter walk/run (10-MWR) Velocity | Baseline, Week 96
Change From Baseline in the North Star Ambulatory Assessment (NSAA) Total Score at Week 96 | Baseline, Week 96
  The NSAA is a clinician administered scale that rates the participant's performance on various functional activities. During this assessment, participants will be asked to perform 17 different functional activities, including a 10 meter walk/run, rising from a sit to standing, standing on 1 leg, climbing a box step, descending a box step, rising from lying to sitting, rising from the floor, lifting the head, standing on heels, and jumping. Participants will be graded as follows: 2 = achieves goal without any assistance; 1 = modified method but achieves goal independent of physical assistance from another person; and 0 = unable to achieve goal independently. NSAA Total Score ranges from 0 to 34, with a score of 34 implying normal function.
Change from Baseline in Dystrophin Protein Levels Determined by Western Blot at Weeks 48 or 96 | Baseline, Week 48 or Week 96
Change from Baseline in Dystrophin Intensity Levels Determined by Immunohistochemistry (IHC) at Weeks 48 or 96 | Baseline, Week 48 or Week 96

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (76):
- United States (23):
  - Neuromuscular Research Center, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - David Geffen School of Medicine, UCLA, Los Angeles, California
  - Rady Children's Hospital San Diego/ UCSD, San Diego, California
  - Stanford University School of Medicine/Medical Center, Stanford, California
  - University of Florida, Gainesville, Florida
  - NW Florida Clinical Research Group, LLC, Gulf Breeze, Florida
  - Center for Integrative Rare Disease Research (CIRDR), Atlanta, Georgia
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - University of Kansas, Medical Center, Kansas City, Kansas
  - Boston Children's Hospital, Boston, Massachusetts
  - St. Louis Children's Hospital, St Louis, Missouri
  - Las Vegas Clinic, Las Vegas, Nevada
  - University of Rochester Clinical Research Center, Rochester, New York
  - Cincinnati Children's Hospital Medical Center (CCHMC), Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Shriners Hospital for Children, Portland, Oregon
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Children's Medical Center Dallas, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- DOM Centro de Reumatologia, Buenos Aires, Argentina
- Australia (3):
  - Royal Children's Hospital Melbourne, Parkville, Victoria
  - Queensland Children's Hospital, South Brisbane
  - Children's Hospital at Westmead, Westmead
- Belgium (3):
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Leuven, Leuven
  - CHR de la Citadelle, Liège
- University Multiprofile Hospital for Active Treatment Aleksandrovska EAD, Sofia, Sofia-Grad, Bulgaria
- Canada (4):
  - Alberta Childrens Hospital, Calgary, Alberta
  - Children's and Women's Health Centre of British Columbia, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
- Czechia (2):
  - University Hospital Brno, Brno
  - Fakultni nemocnice v Motole, Prague
- Rigshospitalet Copenhagen University Hospital, København Ø, Denmark
- France (3):
  - Hôpital Des Enfants, Toulouse, Haute-Garonne
  - Reference Centre for Neuromuscular Diseases, Nantes
  - Hôpital Armand Trousseau, Paris
- Germany (4):
  - LMU Klinikum der Universität, München, Bavaria
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Essen, Essen
  - University Hospital Freiburg, Freiburg im Breisgau
- Greece (2):
  - IASO Children's Hospital, Marousi
  - Ippokratio General Hospital of Thessaloniki, Thessaloniki
- Semmelweis Egyetem Genomikai Medicina és Ritka Betegsegek Intezete, Budapest, Hungary
- India (2):
  - Royal Instituite of Child Neurosciences, Ahmedabad, Gujarat
  - Deenanth Mangeshkar Hospital, Pune, Maharashtra
- The Children's University Hospital, Dublin, Ireland
- Schneider Children's Medical Center of Israel, Petah Tikvah, Israel
- Italy (5):
  - Azienda Ospedaliero-Universitaria di Ferrara - Arcispedale Sant' Anna, Ferrara
  - Istituto Giannina Gaslini, Genoa
  - Az Ospedaliera Universitaria Policlinico G Martino, Messina
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Policlinico Universitario A Gemelli, Rome
- Mexico (2):
  - Neurociencias Estudios Clínicos S.C, Culiacán
  - Instituto de Investigaciones Clínicas para la Salud A.C, Durango
- Poland (2):
  - Samodzielny Publiczny Centralny Szpital Kliniczny, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk
- Russia (2):
  - Federal state budget educational institution of higher education "Russian national research medical university n.a. N.I. Pirogov" of Ministry of healthcare of Russian Federation, Moscow
  - State Autonomous Healthcare Institution of Sverdlovsk Region Children's Clinical Hospital No. 9 City of Ekaterinburg, Yekaterinburg
- Clinic for Neurology and Psychiatry for Children and Youth, Belgrade, Serbia
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (3):
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Drottning Silvias Barn Och Ungdomssjukhus, Gothenburg, Sweden
- United Kingdom (6):
  - Royal Hospital for Children (Glasgow), Glasgow
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Alder Hey Childrens Hospital, Liverpool
  - Great Ormond Street Hospital (GOSH), London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vandekerckhove I, Hanssen B, Peeters N, Dewit T, De Beukelaer N, Van den Hauwe M, De Waele L, Van Campenhout A, De Groote F, Desloovere K. Anthropometric-related percentile curves for muscle size and strength of lower limb muscles of typically developing children. J Anat. 2025 Aug;247(2):348-362. doi: 10.1111/joa.14241. Epub 2025 Mar 17. PMID 40098309
- [Derived] Wagner KR, Kuntz NL, Koenig E, East L, Upadhyay S, Han B, Shieh PB. Safety, tolerability, and pharmacokinetics of casimersen in patients with Duchenne muscular dystrophy amenable to exon 45 skipping: A randomized, double-blind, placebo-controlled, dose-titration trial. Muscle Nerve. 2021 Sep;64(3):285-292. doi: 10.1002/mus.27347. Epub 2021 Jun 29. PMID 34105177